CLINICAL TRIAL: NCT01909024
Title: A Randomised Controlled Trial Investigating The Use Of Pelvic Vein Embolisation To Reduce Recurrent Varicose Veins Of The Legs In Women With Recurrent Varicose Veins And Associated Pelvic Venous Reflux.
Brief Title: Pelvic Embolisation to Reduce Recurrent Varicose Veins - Recurrent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Whiteley Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT23013
Record Dates: First submitted 2013-07-02; First posted 2013-07-26 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Varicose Veins; Venous Reflux; Pelvic Congestion Syndrome
Keywords: Randomised controlled trial; Endovenous laser treatment; Transjugular coil embolisation
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- embolisation of pelvic veins & treatment of leg varicose veins (Experimental): transjugular coil embolisation of pelvic veins followed by endovenous treatment of leg recurrent varicose veins
  Interventions: Procedure: Coil embolisation; Procedure: endovenous treatment of leg recurrent varicose veins
- endovenous treatment of leg recurrent varicose veins alone (Active Comparator): endovenous treatment of leg recurrent varicose veins alone
  Interventions: Procedure: endovenous treatment of leg recurrent varicose veins

INTERVENTIONS:
Procedure: Coil embolisation — transjugular coil embolisation of pelvic veins
  Arms: embolisation of pelvic veins & treatment of leg varicose veins
Procedure: endovenous treatment of leg recurrent varicose veins — endovenous treatment of leg recurrent varicose veins

SUMMARY:
The aim of this study is to identify whether the treatment of pelvic venous reflux (pelvic embolisation) in females with recurrent leg varicose veins, who have a proven contribution to their leg varicose veins from pelvic venous reflux, have a reduction in future recurrence after endovenous laser treatment for recurrent varicose veins in the legs.

DETAILED DESCRIPTION:
Varicose veins of the legs effect between 20 and 40% of the adult population in the UK. Approximately 100,000 operations performed per year for varicose veins, although it is unknown how many of these are for recurrent varicose veins. Failure to treat varicose veins results in 10 to 20% of patients deteriorating to skin damage or leg ulceration. Recurrence rates following surgery vary and have been reported up to 70% at 10 years. Recurrence causes an increased cost as well as an increase in the patient's healthcare requirements.

The commonest causes of recurrence are reported to be:

* neovascularisation (new vessel growth after treatment)
* missing veins at the initial operation
* perforator vein incompetence
* de novo reflux due to normal deterioration with age

Recent studies have shown that leg varicose veins can be caused by pelvic venous reflux and that pelvic venous reflux is a cause of recurrent varicose veins. Previous published work from our own unit has shown that approximately 20% of women who present with varicose veins of the legs and who have had children previously have pelvic venous reflux on duplex ultrasound. Such pelvic venous reflux contributes to the venous reflux in the legs, causing the varicose veins. Furthermore, a recent retrospective study from our own unit has suggested that failure to treat pelvic venous reflux before treating leg varicose veins is a major cause of recurrent varicose veins in up to a quarter of women.

However, despite this circumstantial evidence, there is no evidence to prove whether the treatment of pelvic venous reflux confers any advantage on these patients in terms of reduction in future recurrence of their varicose veins, following treatment.

The treatment of pelvic venous reflux is currently by coil embolisation of the veins under x-ray control. This procedure clearly has an additional cost over and above that of treating the leg varicose veins alone. Therefore it is essential to know whether the treatment of the pelvic veins in these patients has any effect in reducing future recurrence of leg varicose veins.

To examine the benefits of coil embolisation, female patients presenting with recurrent leg varicose veins with a duplex proven contribution from pelvic venous reflux will be randomised to:

1. transjugular coil embolisation of pelvic veins followed by endovenous treatment of leg recurrent varicose veins

   or
2. endovenous treatment of leg recurrent varicose veins alone

The impact of demographic factors, the severity of patient's symptoms(Aberdeen questionnaire, CEAP and VCCS scores)and treatment history will be explored, in addition to the type of treatment received.

Patients will be followed up at six weeks, six months, one year, two years, three years, four years and five years.

Outcome measures will include quality-of-life scoring (CIVIQ), symptom severity measures (Aberdeen questionnaire, CEAP and VCCS scores), patient satisfaction with treatment and clinical examination including clinical photographs and duplex ultrasonography.

The source of any recurrence will be classified through the use of duplex ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Females presenting with recurrent varicose veins in one or both legs with ultrasound proven pelvic venous reflux in at least one pelvic venous trunk communicating with the leg varicose veins
* Duplex proven reflux in the superficial venous system of the leg
* Over 18 years old
* Able to understand and give consent
* Willing to attend for follow-up over the five years

Exclusion Criteria:

* Pelvic venous reflux does not communicate with the varicose veins to be treated in the legs
* If pelvic venous reflux communicates and contributes to varicose veins in one leg but not the other, only the leg with a pelvic venous contribution will be entered into the study
* Currently pregnant or plans for pregnancy within the next five years
* Under 18 years of age
* Unable to understand all give consent
* Any vascular malformation of the pelvis all the legs apart from that diagnosed as venous reflux disease
* Any medical condition likely to cause death or serious ill-health within the next five years Any deep venous obstruction or reflux

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2013-07; Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in recurrent varicose veins or venus reflux | 6 weeks, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years post surgery
  Does the patient have recurrence?
  Recurrent varicose veins will be divided into:
  * Clinically insignificant (thread veins, reticular veins or varicose veins less than 3 mm in diameter)
  * Significant (varicose veins greater than 3 mm in diameter, varicose veins associated with thrombophlebitis, or skin changes such as venous eczema, red skin or Brown skin overlying the veins)

SECONDARY OUTCOMES:
Quality of life | 6 weeks post surgery, 6 months post surgery, 1 year post surgery, 2 years post surgery, 3 years post surgery, 4 years post surgery, 5 years post surgery
  Participants will complete the Chronic Venous Insufficiency Questionnaire (CIVIQ)
  The CIVIQ comprises 20 questions in four quality-of-life domains: physical, psychological, social, and pain.
Patient satisfaction | 6 weeks post surgery, 6 months post surgery, 1 year post surgery, 2 years post surgery, 3 years post surgery, 4 years post surgery, 5 years post surgery
  Participants will complete a visual analogue scale, from 0 (completely dissatisfied) to 10 (completely satisfied) to indicate their level of satisfaction with the treatment that they have received.
Symptom severity | 6 weeks post surgery, 6 months post surgery, 1 year post surgery, 2 years post surgery, 3 years post surgery, 4 years post surgery, 5 years post surgery
  Participants will complete the Aberdeen questionnaire to assess the severity and impact of their varicose veins on their lives.
  Duplex ultrasound, the CEAP and VCCS will also be used to assess the severity of symptoms.
Source of recurrence | 6 weeks post surgery, 6 months post surgery, 1 year post surgery, 2 years post surgery, 3 years post surgery, 4 years post surgery, 5 years post surgery
  Duplex ultrasound will be used to identify the source of any recurrent varicose veins, enabling classification into:
  recurrence due to pelvic venous incompetence recurrence of leg varicose veins due to failure of surgery recurrence of leg varicose veins due to de novo reflux

OTHER OUTCOMES:
Adverse events | 6 weeks post surgery, 6 months post surgery, 1 year post surgery, 2 years post surgery, 3 years post surgery, 4 years post surgery, 5 years post surgery
  Incidences of thrombophlebitis and deep vein thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Whiteley, Professor, Principal Investigator — The Whiteley Clinic
Locations (2):
- United Kingdom (2):
  - The Whiteley Clinic, Guildford
  - The Imaging Clinic, Guildford